CLINICAL TRIAL: NCT04639505
Title: Predictive Value of New AMH Test Method for Ovarian Response in Patients With IVF/ICSI
Brief Title: Predictive Value of New AMH Test Method for Ovarian Response
Status: Completed | Type: Observational
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Other Study IDs: P2020004
Record Dates: First submitted 2020-11-11; First posted 2020-11-20 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Infertility; AMH
MeSH Terms: conditions — Infertility | interventions — Luminescence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ELISA: ELISA kit detecting the serum AMH level
  Interventions: Diagnostic Test: ELISA
- Chemiluminescence: CLIA method detecting the serum AMH level
  Interventions: Diagnostic Test: Chemiluminescence

INTERVENTIONS:
Diagnostic Test: ELISA — ELISA kit detecting the serum AMH level
  Other Names: experimental group
  Groups: ELISA
Diagnostic Test: Chemiluminescence — CLIA method detecting the serum AMH level
  Other Names: control group
  Groups: Chemiluminescence

SUMMARY:
In China, the incidence of infertility is about 15%, and patients need to use assisted reproductive technology (ART) to obtain pregnancy. It is particularly important to accurately predict the patient's ovarian response before initiating controlled ovulation hyperstimulation (COH). At present, the commonly used AMH detection method is enzyme-linked immunoassay (ELISA), and it has obtained the normal reference range for ovarian response. In recent years, with the development of detection technology, chemiluminescence immunoassay（CLIA） detection reagents have been successively used for the detection of AMH. However, there are few studies on the comparison of these two detection methods. The predictive value of the new method on ovarian response was lack. Therefore, by comparing the two methods of ELISA and CLIA detection of AMH levels in this study, the predictive value of poor ovarian response (the number of retrieved oocyte ≤ 3) and high response (the number of retrieved oocyte ≥ 15) in IVF/ICSI stimulation cycle was analyzed. In order to provide more reference basis for individualized COH, the AMH cutoff value of low and high ovarian response by the new method predicts was analyzed. At the same time, the prediction value of the two methods is compared to determine whether the new CLIA is suitable for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* The first IVF/ICSI COH cycle;
* the causes of infertility :fallopian tube factors and/or male factors;

Exclusion Criteria:

* Endometriosis;
* PCOS;
* Adenomyosis;
* PGT cycle because of the female chromosome abnormality or genetic abnormality;
* FET cycle;
* Malignant tumor patient.

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: infertility females
Sampling Method: Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
the AMH（CLIA） cutoff value of low and high ovarian response | the day of oocytes retrieved，about three months after AMH test
  the poor ovarian response :the number of retrieved oocyte ≤ 3,the high ovarian response :the number of retrieved oocyte ≥ 15

SECONDARY OUTCOMES:
Number of oocytes retrieved | 34-36 hours after hCG trigger，about three months after AMH test
  the number of oocytes retrieved after hCG trigger
the serum AMH level | any day of the menstrual cycle, about three months after study starting
  anti-muller hormone

CONTACTS AND LOCATIONS:
Overall Officials: Fei Gong, PhD, Principal Investigator — Reproductive & Genetic Hospital of CITIC-Xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China